CLINICAL TRIAL: NCT07356427
Title: Effects of Virtual Reality Tennis Training on Self-Efficacy, Flow Experience, Embodied Cognition, and Intention to Use Among Chinese University Tennis Players: A Randomized Controlled Trial
Brief Title: VR Tennis Training Effects on Psychological Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, ROHAYU BINTI HAMI, Doctoral, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: USM/JEPeM/PP/25030255
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sports Performance; Psychological Adaptation
Keywords: Virtual Reality; Tennis; Flow Experience; Embodied Cognition; Technology Acceptance; Sports Psychology; Self-Efficacy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the VR tennis training group or the traditional tennis training control group in a 1:1 ratio, with both groups receiving training concurrently over the 8-week intervention period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who administered questionnaires and collected data were blinded to participant group allocation. Due to the nature of the interventions, participants and training providers could not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Tennis Training (Experimental): Participants received 8 weeks of immersive VR tennis training using Meta Quest 2 headsets. Training sessions were conducted twice weekly, each lasting 60 minutes (16 sessions total). Sessions included warm-up in virtual environment (10 min), technical skill practice (25 min), tactical decision-making scenarios (20 min), and cool-down (5 min).
  Interventions: Behavioral: Traditional Tennis Training
- Traditional Tennis Training (Active Comparator): Participants received 8 weeks of traditional tennis training matched for frequency (twice weekly), duration (60 minutes/session), and content structure. Sessions included physical warm-up (10 min), technical skill drills (25 min), point play and match simulation (20 min), and cool-down (5 min).
  Interventions: Behavioral: Virtual Reality Tennis Training

INTERVENTIONS:
Behavioral: Virtual Reality Tennis Training — Immersive VR tennis training using Meta Quest 2 head-mounted displays. The VR system provided real-time feedback on stroke mechanics, ball trajectory, and court positioning. Training included progressive difficulty adjustment based on individual performance. Participants practiced forehand, backhand, serve techniques, and tactical decision-making against virtual opponents.
  Arms: Traditional Tennis Training
Behavioral: Traditional Tennis Training — Standard tennis training delivered by qualified coaches on regular tennis courts. Training included ball feeding machines, partner practice, and coach-led instruction for technical skills, as well as competitive rallies for tactical application.
  Arms: Virtual Reality Tennis Training

SUMMARY:
This randomized controlled trial examined the effects of an 8-week virtual reality (VR) tennis training intervention on psychological outcomes among Chinese university tennis players.

A total of 180 participants were randomly assigned to either a VR training group (n=90) using Meta Quest 2 headsets or a traditional training control group (n=90). The VR group received immersive tennis training twice weekly for 60 minutes per session, while the control group received equivalent traditional coaching.

Primary outcomes included self-efficacy, flow experience, embodied cognition, and intention to use, measured at baseline and post-intervention. Secondary analyses examined whether self-efficacy and flow experience mediated the relationship between VR training and intention to use.

The study aimed to provide evidence for the effectiveness of VR technology in sports training and to elucidate the psychological mechanisms underlying VR training benefits.

DETAILED DESCRIPTION:
Background:

Virtual reality (VR) technology has emerged as a promising tool for sports training, offering immersive environments that simulate real-world athletic scenarios. Tennis represents an ideal sport for VR training applications due to its technical complexity, spatial demands, and the importance of anticipatory skills. Despite growing adoption of VR in sports contexts, the psychological mechanisms underlying VR training effectiveness remain insufficiently understood.

Theoretical Framework:

This study was grounded in four theoretical perspectives: (1) Bandura's Self-Efficacy Theory, proposing that VR training enhances confidence through mastery experiences; (2) Csikszentmihalyi's Flow Theory, suggesting VR environments facilitate optimal psychological states; (3) Embodied Cognition Theory, emphasizing that cognitive processes are rooted in bodily interactions; and (4) the Technology Acceptance Model, providing a framework for understanding intention to use technology.

Objectives:

Primary objectives were to determine whether VR tennis training produces greater improvements in self-efficacy, flow experience, embodied cognition, and intention to use compared to traditional training. Secondary objectives investigated whether self-efficacy and flow experience mediate the effect of VR training on intention to use.

Methods:

A parallel-group, single-blind randomized controlled trial was conducted at Hezhou University, Guangxi, China. Eligible participants were undergraduate students aged 18-26 years enrolled in Physical Education or Sports Science programs with at least two semesters of tennis instruction. Participants were randomly assigned using computer-generated random numbers with stratification by sex and year of study.

Intervention:

The VR group received 8 weeks of immersive tennis training using Meta Quest 2 head-mounted displays (2 sessions/week, 60 minutes/session, 16 sessions total). Training included warm-up in virtual environment (10 min), technical skill practice (25 min), tactical decision-making scenarios (20 min), and cool-down (5 min). The control group received matched traditional tennis training with the same frequency, duration, and content structure.

Outcome Measures:

Self-efficacy was measured using an 8-item scale adapted from Bandura (2006). Flow experience was assessed using a 10-item scale based on Csikszentmihalyi (1990). Embodied cognition was measured using an 8-item scale adapted from presence questionnaires. Intention to use was assessed with a 6-item scale adapted from the Technology Acceptance Model. Sport motivation (SMS-II) was measured as a covariate.

Statistical Analysis:

Between-group differences were examined using analysis of covariance (ANCOVA) controlling for baseline scores and sport motivation. Effect sizes were calculated as Hedges' g. Parallel mediation analysis was conducted using the PROCESS macro with bias-corrected bootstrap confidence intervals (10,000 samples).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students aged 18-26 years
* Enrolled in Physical Education or Sports Science programs at Hezhou University
* Completed at least two semesters of formal tennis instruction
* Basic tennis proficiency (able to perform forehand, backhand, and serve)
* Willing to participate in the 8-week training program
* Able to provide written informed consent

Exclusion Criteria:

* Visual impairments that could not be corrected and would preclude VR headset use
* History of photosensitive epilepsy or seizure disorders
* Vestibular disorders or severe motion sickness
* Current participation in competitive tennis programs at regional or higher levels
* Prior experience with VR-based sports training systems
* Any musculoskeletal injury preventing full participation in tennis training

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | Baseline and 8 weeks (post-intervention)
  Tennis-specific self-efficacy measured using an 8-item scale adapted from Bandura (2006). Items assess confidence in performing tennis skills and managing competitive situations. Responses on 5-point Likert scale (1=Strongly Disagree to 5=Strongly Agree). Higher scores indicate greater self-efficacy. Score range: 1-5.
Flow Experience | Baseline and 8 weeks (post-intervention)
  Flow during training measured using a 10-item scale based on Csikszentmihalyi (1990). Items assess challenge-skill balance, concentration, sense of control, and intrinsic enjoyment. Responses on 5-point Likert scale. Higher scores indicate greater flow experience. Score range: 1-5.
Embodied Cognition | Baseline and 8 weeks (post-intervention)
  Embodied cognition during training measured using an 8-item scale adapted from presence questionnaires (Wilson 2002; Gonzalez-Franco 2018). Items assess sense of presence, body ownership, and sense of agency. Responses on 5-point Likert scale. Higher scores indicate greater embodied cognition. Score range: 1-5.
Intention to Use | Baseline and 8 weeks (post-intervention)
  Intention to continue using the training method measured using a 6-item scale adapted from the Technology Acceptance Model (Davis 1989). Items assess willingness to use, recommend, and prefer the training method. Responses on 5-point Likert scale. Higher scores indicate greater intention to use. Score range: 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, PhD Candidate, Principal Investigator — Advanced Medical and Dental Institute, Universiti Sains Malaysia; Rohayu Hami, PhD, Study Director — Advanced Medical and Dental Institute, Universiti Sains Malaysia
Locations (1):
- Hezhou University, Hezhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No
This study was conducted as part of a doctoral dissertation. The informed consent obtained from participants did not include provisions for sharing individual-level data with external researchers.